CLINICAL TRIAL: NCT03998839
Title: Monitoring of Markers of Sulfadoxine-pyrimethamine (SP) Resistance in the Implementation Countries of TIPTOP Project
Brief Title: TIPTOP Sulfadoxine-pyrimethamine (SP) Drug Resistance Study
Acronym: TIPTOP-DRS
Status: Completed | Type: Observational
Sponsor: Jhpiego (Other)
Collaborators: Barcelona Institute for Global Health (Other)
Responsible Party: Sponsor
Other Study IDs: TIPTOP_DRS_2019
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Malaria in Pregnancy
Keywords: drug resistance; Sulfadoxine-pyrimethamine

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — During the surveys, blood samples will be collected onto filter papers (dried blood spots). The surveys will be undertaken in the intervention area (the initial area of implementation of C-IPTp) and one control area (with no C-IPTp) in each country (Figure 1). C-IPTp-SP delivery in the area of initial implementation will start immediately after baseline surveys and sample collection. The sample collection will be performed in four selected first level of care health facilities in the intervention area and four health facilities in the control area.
  The key markers to be monitored are dihydrofolate reductase (dhfr) triple mutation (codon 108, 51 and 59) together with triple P. falciparum dihydropteorate synthetase (dhps) mutations at codons 431, 437, 540, 581 and 613.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intervention: Children tested will live within an area targeted for community IPTp distribution for pregnant women.
  Interventions: Other: Community distribution of Sulfadoxine-pyrimethamine (SP)
- Control: Children tested will live within an area NOT targeted for C-IPTp, but will live in an area nearby.

INTERVENTIONS:
Other: Community distribution of Sulfadoxine-pyrimethamine (SP) — Community health workers will distribute SP to pregnant women, targeting at least three times during pregnancy.
  Other Names: C-IPTp-SP
  Groups: Intervention

SUMMARY:
The main objective of this study is to monitor SP resistance via molecular markers in the context of the TIPTOP project implementation of community distributed SP for women during pregnancy.

The specific objective is to detect trends over time in the proportion of symptomatic children with a positive rapid diagnostic test (RDT) residing in the areas where C-IPTp is implemented who carry parasites with dhfr/dhps mutations compared to those in control areas with no community SP distribution.

DETAILED DESCRIPTION:
The TIPTOP (Transforming Intermittent Preventive Treatment for Optimal Pregnancy) project will explore an alternative innovative approach to antenatal care (ANC) facilities or clinic for the delivery of IPTp-SP. It will sustain and scale up a community-based delivery system to be implemented in addition to the traditional ANC clinic-based delivery system with the aim of expanding coverage of IPTp-SP. The innovative approach, called community IPTp (C-IPTp-SP), will be implemented in four sub-Saharan African countries: Nigeria, Democratic Republic of Congo (DRC), Madagascar and Mozambique. TIPTOP will use community health workers (CHWs) as a delivery channel to increase coverage of IPTp-SP to a minimum of 50% in project areas to prevent malaria in pregnancy (MiP). It is expected that this will lead to a substantial increase in the consumption of SP, not supervised by professional health workers. To address the concern that this may lead to an increase in the accumulation of mutations in dihydrofolate reductase (dhfr) and dihydropteroate synthetase (dhps) that could lead to an increase of the parasite resistance to SP, TIPTOP will monitor the prevalence of molecular markers of SP resistance in the population at three times during the project: at baseline, midline - following approximately 18 months of implementation - and endline - after 3 years of implementation. Providing evidence on the effects on SP resistance of C-IPTp is important for decision-making as to whether C-IPTp can be recommended as an additional channel for IPTp delivery or if the use of an alternative drug for IPTp should be considered. Moreover, it is expected that the SP resistance monitoring will also help to mitigate the risk of perceiving SP as a failed drug negatively affecting demand for quality-assured (QA) SP for IPTp (risk management). C-IPTp will be implemented in each country initially in a "test" area (Phase I) and later expanded to two additional areas (Table 1). All areas have been selected purposefully. Trends of SP resistance will be monitored in the initial "test" area, with C-IPTp, and in a neighbouring area with similar epidemiologic characteristics but with no C-IPTp (control area). A health facility-based, cross-sectional survey will be conducted before project implementation (baseline), after 18 months of intervention (midline) and after three years of intervention (endline) to measure the prevalence of molecular markers associated with resistance to SP in symptomatic children under five years of age with a positive RDT attending selected health facilities in the intervention and control areas. Monitoring the prevalence of alleles associated with resistance to drugs is, by standard protocol, done by collecting samples from symptomatic children with evidence of infection. The rationale for this is that any over- or misuse of drug in any sub-population, including pregnant women, may select parasites strains resistant to SP and that those strains are then transferred by mosquitos to the general population and most easily detected in children.

During the surveys, blood samples will be collected onto filter papers (dried blood spots). The surveys will be undertaken in the intervention area (the initial area of implementation of C-IPTp) and one control area (with no C-IPTp) in each country (Figure 1). C-IPTp-SP delivery in the area of initial implementation will start immediately after baseline surveys and sample collection. The sample collection will be performed in four selected first level of care health facilities in the intervention area and four health facilities in the control area.

ELIGIBILITY:
Inclusion Criteria:

* • Children under five years of age.

  * Being resident in the project area at the time of the survey.
  * Clinical signs and symptoms suggestive of malaria infection: fever (axillary temperature ≥37.5ºC) or history of fever in the preceding 24 hours.

Exclusion Criteria:

* Not willing to provide informed consent
* Signs or symptoms of severe malaria

Ages: 0 Years to 5 Years | Sex: All
Age Groups: Child
Study Population: Study population will be children under five years of age attending the selected health facilities in the intervention and control areas.
Sampling Method: Non-Probability Sample
Enrollment: 7200 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
change in prevalence of molecular markers associated with SP resistance at 36 months | baseline to endline (approximately 36 months later)
  change in prevalence of molecular markers associated with SP resistance (codons 108, 51 and 59 in dhfr and 437, 540 and 581 in dhps) in blood samples collected from symptomatic children under five years with a positive RDT attending the selected health facilities at 36 months (baseline to endline)
change in prevalence of molecular markers associated with SP resistance at 18 months | baseline to midline (approximately 18 months later)
  change in prevalence of molecular markers associated with SP resistance (codons 108, 51 and 59 in dhfr and 437, 540 and 581 in dhps) in blood samples collected from symptomatic children under five years with a positive RDT attending the selected health facilities. from baseline to midline (18 months)

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Roman, MA, Study Director — Jhpiego
Locations (4):
- Kenge District, Community Setting, Kenge, Kwango, Democratic Republic of the Congo
- Mananjary District, Community Setting, Mananjary, Fianarantsoa, Madagascar
- Nhamatanda District, Community Setting, Nhamatanda, Sofala, Mozambique
- Ohaukwu District, Community Setting, Ohaukwu, Ebonyi State, Nigeria

IPD SHARING:
Plan to Share IPD: No
At this time there is no plan to share the individual-level data with other researchers.